CLINICAL TRIAL: NCT06812884
Title: Effects of Education Given to Retrograde Intrarenal Surgery Patients With Mobile Application on Anxiety, Fear of Surgery, Pain, Analgesic Consumption, Length of Hospital Stay, Complication Development, Readmission and Hospitalization
Brief Title: Effects of Education Given to RIRS With Mobile Application on Anxiety, Fear of Surgery, Pain, Analgesic Consumption, Length of Hospital Stay, Complication Development, Readmission and Hospitalization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Collaborators: Mersin University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Dr, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: TU-BOZKUL-011
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Retrograde Intrarenal Surgery
Keywords: Mobile application; Patient education; Nursing; Patient outcome
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The assignment of the patients included in the study to the groups will be carried out by the researcher (SY), who is not involved in the data collection process, with the simple randomization method of random numbers table. The https://www.randomizer.org/ website will be utilized in the table formation. When the patient who will undergo RIRC comes to the urology clinic, researchers GB and MB will evaluate the patients in terms of inclusion criteria. When the patient meets the inclusion criteria and signs the informed consent form, GB will inform the researcher SY and SY will inform GB which group the patient will be assigned to. In this way, all researchers, patients, patients' relatives and clinic staff other than the HC will be blinded to group assignment. In order to prevent bias in statistical analyses, the data of the patients whose data collection process is completed will be coded as G1, G2 and G3 by the researcher GAU without specifying the group name and entered into the data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Mobile application group (Experimental): "Introductory Information Form", 'State Anxiety Scale', and 'Surgical Fear Scale' will be applied to all patients before surgical intervention. "State Anxiety Scale" and 'Surgical Fear Scale' will be administered both before and after the trainings in the preoperative period. The trainings and the scales to be filled out before surgery will be carried out when the patient is admitted to the clinic for surgery. The group to be trained with the mobile application will be introduced to the application and the application will be downloaded to their phones, tablets or computers. After the surgical intervention, "VAS" and "Analgesic Consumption Monitoring Form" will be applied to all patients. Patients' pain will be evaluated with VAS when they come to the postoperative room, postoperative 6th hour and postoperative 12th hour. The amount of analgesia consumed by the patients within 24 hours postoperatively will be recorded in the Analgesia Consumption Form. The duration of hospital stay wi
  Interventions: Other: Education
- Control group (No Intervention): Patients in the control group will receive the routine information provided in the clinic. All patients will be administered "Descriptive Information Form", "State Anxiety Scale", and "Surgical Fear Scale" before surgical intervention. "State Anxiety Scale" and 'Surgical Fear Scale' will be administered both before and at the end of the briefing in the preoperative period. After the surgical intervention, "VAS" and "Analgesic Consumption Monitoring Form" will be applied to all patients. The pain of the patients will be evaluated with VAS when they come to the postoperative room, at the 6th postoperative hour and at the 12th postoperative hour. The amount of analgesia consumed by the patients within 24 hours postoperatively will be recorded in the Analgesia Consumption Form. The duration of hospital stay will be recorded on the "Patient Follow-up Form" on the day of discharge.

INTERVENTIONS:
Other: Education — The mobile application will be introduced to the group to be trained and the application will be downloaded to their phones, tablets or computers.
  Arms: Experimental: Mobile application group

SUMMARY:
The aim of this study was to determine the effect of the education to be given with a mobile application to be developed for RIRC patients on preoperative anxiety, fear of surgery, postoperative pain level, analgesic consumption, length of hospital stay, development of complications in the first month, readmission and number of hospitalizations. The study was planned as a prospective, two-arm (1:1), randomized controlled trial. The study will be conducted with 68 patients in the urology clinic of a university hospital. Patients will be randomly assigned to the control group and the mobile application training group.. Descriptive Information Form, Visual Analog Scale (VAS), Analgesic Consumption Monitoring Form, State Anxiety Scale, Surgical Fear Scale and Patient Monitoring Form will be used to collect the data. "Introductory Information Form", 'State Anxiety Scale', and 'Surgical Fear Scale' will be applied to all patients before surgical intervention. "State Anxiety Scale" and 'Surgical Fear Scale' will be administered both before and at the end of the trainings in the preoperative period. Trainings and preoperative scales to be completed will be carried out when the patient is admitted to the clinic for surgery. The group to be trained with the mobile application will be introduced to the application and the application will be downloaded to their phones, tablets or computers. Then, the questions of the patients regarding the mobile application will be answered. Patients in the control group will receive routine information in the clinic. After the surgical intervention, "VAS" and "Analgesic Consumption Monitoring Form" will be applied to all patients. The pain of the patients will be evaluated with VAS when they come to the postoperative room, at the 6th postoperative hour and at the 12th postoperative hour. The amount of analgesia consumed by the patients within 24 hours postoperatively will be recorded in the Analgesia Consumption Form. The duration of hospital stay will be recorded on the "Patient Follow-up Form" on the day of discharge. Patients who underwent RIRC will be called by the investigators one month later and their complication development status, hospitalization/ rehospitalization status will be learned and recorded in the "Patient Follow-up Form".

DETAILED DESCRIPTION:
The aim of this study was to determine the effect of the education to be given with a mobile application to be developed for RIRC patients on preoperative anxiety, fear of surgery, postoperative pain level, analgesic consumption, length of hospital stay, development of complications in the first month, readmission and number of hospitalizations. The study was planned as a prospective, two-arm (1:1), randomized controlled trial. The study will be conducted with 68 patients in the urology clinic of a university hospital. Patients will be randomly assigned to the control group and the mobile application training group. Patients in the mobile application group will be trained with the mobile application, while patients in the control group will only receive routine care in the clinic. Patients assigned to the mobile application group will be introduced to the education to be given with the mobile application and the application will be downloaded to their phones/tablets. Descriptive Information Form, Visual Analog Scale (VAS), Analgesic Consumption Monitoring Form, State Anxiety Scale, Surgical Fear Scale and Patient Monitoring Form will be used to collect the data. "Introductory Information Form", 'State Anxiety Scale', and 'Surgical Fear Scale' will be applied to all patients before surgical intervention. "State Anxiety Scale" and 'Surgical Fear Scale' will be administered both before and at the end of the trainings in the preoperative period. Trainings and preoperative scales to be completed will be carried out when the patient is admitted to the clinic for surgery. The group to be trained with the mobile application will be introduced to the application and the application will be downloaded to their phones, tablets or computers. Then, the questions of the patients regarding the mobile application will be answered. Patients in the control group will receive routine information in the clinic. After the surgical intervention, "VAS" and "Analgesic Consumption Monitoring Form" will be applied to all patients. The pain of the patients will be evaluated with VAS when they come to the postoperative room, at the 6th postoperative hour and at the 12th postoperative hour. The amount of analgesia consumed by the patients within 24 hours postoperatively will be recorded in the Analgesia Consumption Form. The duration of hospital stay will be recorded on the "Patient Follow-up Form" on the day of discharge. Patients who underwent RIRC will be called by the investigators one month later and their complication development status, hospitalization/ rehospitalization status will be learned and recorded in the "Patient Follow-up Form".

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Elective RIRC planned,
* Conscious, oriented and cooperative,
* Written permission to participate in the study was obtained,
* Who speaks and understands Turkish,
* Literate,
* Not visually or hearing impaired,
* Not mentally disturbed,
* The person or caregiver has an android phone or tablet,
* Using an android phone or tablet for at least a year,
* Patients who state that they do not have any disability related to the use of technology will be included in the study.

Exclusion Criteria:

* Emergency RIRC planned,

  * Under 18 years old,
  * Refused to participate in the research,
  * Who doesn't speak Turkish,
  * Illiterate,
  * Undergoing other surgical interventions in conjunction with RIRC,
  * Visually or hearing impaired,
  * Neither they nor their caregiver has an android phone or tablet
  * Have used a smartphone or tablet for less than one year,
  * Patients who state that they have a disability related to the use of technology will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
Pain score | 6 months
  Visual Analog Scale: It is a scale that provides a subjective assessment of pain on a horizontal or vertical line from 0 (no pain at all)-10 (very severe pain) to evaluate the level of pain (Wewers and Lowe, 1990).
Analgesic Consumption | 6 months
  Analgesic Consumption Monitoring Form : In this form, the analgesics consumed by the patients in the first 24 hours after surgical intervention and their amounts will be recorded.
Anxiety | 6 months
  Description: The State Anxiety Scale : In this study, the DAQ, which is structured to measure momentary feelings, was used. Its Turkish validity and reliability was conducted by Öner and Le Compte in 1983. The DAQ consists of 20 questions on a four-point Likert scale. The statements in the DAQ are evaluated as not at all (1), a little (2), a lot (3) and completely (4). In this section, the statements are divided into direct and reversed statements. Inverted statements: 1st, 2nd, 5th, 5th, 8th, 8th, 10th, 11th, 15th, 16th, 19th, 20th items. The total score of the reversed statements is subtracted from the total score of the direct statements and the number 50, which is the invariant value of the DAQ, is added to the value obtained and the DAQ score is calculated. The scale score ranges between 20-80 and an increase in the score indicates an increase in the level of anxiety.
Surgical Fear | 6 months
  Surgical Fear Scale: The Turkish validity and reliability study of the scale was conducted by Bağdigen and Karaman Özlü in 2018. The questionnaire, which consists of eight items, has an 11-point Likert structure ranging from 0 (I am not afraid at all) to 10 (I am very afraid). The questionnaire has two subscales indicating the fear of short-term and long-term consequences of surgery. The subscale score is obtained by summing the scores of the four items in the subscales of the questionnaire. The total score of the questionnaire will be obtained by summing the scores of the two subscales, with a minimum score of 0 and a maximum score of 80. The Cronbach alpha coefficient of the scale was found to be 0.89, 0.86 for the short-term outcomes sub-dimension and 0.87 for the long-term outcomes (Bağdiven & Karaman Özlü, 2016).

SECONDARY OUTCOMES:
Duration of hospital stay | 6 months
  Patient Follow-up Form: This form consists of a chart recording the duration of hospital stay, the development of complications in the first month, the number of readmissions and hospitalizations after RIRC.
Complications | 6 months
  Patient Follow-up Form: This form consists of a chart recording the duration of hospital stay, the development of complications in the first month, the number of readmissions and hospitalizations after RIRC.
Readmissions and hospitilizations | 6 months
  Patient Follow-up Form: This form consists of a chart recording the duration of hospital stay, the development of complications in the first month, the number of readmissions and hospitalizations after RIRC.

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Yüksel, Principal Investigator — Necmettin Erbakan University; Gülay ALTUN UĞRAŞ, Principal Investigator — Mersin University; Murat BOZLU, Principal Investigator — Mersin University
Locations (1):
- Tarsus University, Mersin, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 7. Gerlitz, R. (2017). Barriers and facilitators of preoperative education within Enhanced Recovery after Surgery (ERAS) programs. University of Lethbridge. Faculty of Health Sciences. Master of Nursing
- [Result] Aghamir SMK. Successful retrograde intrarenal surgery (RIRS) for a 2-centimeter stone in a chronic renal failure (CRF) patient. Int J Surg Case Rep. 2021 Oct;87:106375. doi: 10.1016/j.ijscr.2021.106375. Epub 2021 Sep 14. PMID 34534812
- [Result] Abdelmowla, R. A. A., Hussein, A. H., Shahat, A. A., Ahmed, H. A., & Abdelmowla, M. A. A. (2017). Impact of nursing interventions and patients education on quality of life regarding renal stones treated by percutaneous nephrolithotomy. Journal of Nursing Education and Practice, 7(12), 52-63. https://doi.org/10.5430/jnep.v7n12p52